CLINICAL TRIAL: NCT05161793
Title: Telemedicine Continuous Remote Monitoring of Adults With Uncontrolled Diabetes Mellitus
Acronym: TELEMTRRDM
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Anne Peters, Professor, University of Southern California
Other Study IDs: TELE-MONITOR DM
Record Dates: First submitted 2021-12-03; First posted 2021-12-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Continuous Glucose Monitoring; Remote Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CGM-Tele-monitoring Type 1: Tele-CGM-monitoring: Subjects are remotely monitored daily through a continuous glucose monitoring (CGM) system (Libre 2) that communicates via smart phone to a Libreview designed dashboard. Alerts set for: ≥4 hours without CGM signal, ≥2 hours 54-70 mg/dl, and 15 minutes <54 mg/dl. Libreview dashboard automatically emails daily alerts to the Certified Diabetes Care and Education Specialist (CDCES). If alerts occurred, the CDCES performed telemedicine outreach based on type of alert.
  Interventions: Device: Tele-Monitor DM
- CGM-Tele-monitoring Type 2: Tele-CGM-monitoring: Subjects are remotely monitored daily through a continuous glucose monitoring (CGM) system (Libre 2) that communicates via smart phone to a Libreview designed dashboard. Alerts set for: ≥4 hours without CGM signal, ≥2 hours 54-70 mg/dl, and 15 minutes <54 mg/dl. Libreview dashboard automatically emails daily alerts to the Certified Diabetes Care and Education Specialist (CDCES). If alerts occurred, the CDCES performed telemedicine outreach based on type of alert.
  Interventions: Device: Tele-Monitor DM

INTERVENTIONS:
Device: Tele-Monitor DM — Remote monitoring of CGM data to identify, contact, and provide diabetes management for patients who are having episodes of hypoglycemia, hyperglycemia and/or difficulty using their CGM device.

SUMMARY:
The purpose of this single center observational study is to determine the effect of continuous remote continuous glucose monitor (CGM) reporting coupled with a telemedicine intervention (Tele-CGM program) on levels of HbA1C in adults with poorly controlled type 1 or type 2 diabetes. The investigators will follow 200 English and Spanish speaking adults (125 type 2 and 75 type 1 patients) who have an HbA1C >8% over 12 months. The primary analysis will follow the intention-to-treat principle; participants will all be offered the intervention. The primary trial outcome of HbA1c/Glucose Management Indicator (GMI) at 6 and 12 months will be compared from baseline using a linear regression model. The primary independent variable will be the HbA1C from baseline to 6 and 12 months. Patients will serve as their own control. Results will be summarized as group-specific mean, standard deviation (SD) HbA1c, along with a mean treatment difference and 95% confidence interval. Model assumptions including normality and homoscedasticity of residuals will be evaluated; normalizing transformations or rank-based non-parametric procedures will be used as needed. The complete evaluation of HbA1c, including baseline, 6-month and 12 month measurements will be analyzed with mixed effects linear regression, specifying a random participant-level intercept and an unstructured covariance matrix, to accommodate the repeatedly measured data. The secondary trial outcomes of time in range (TIR; CGM glucose levels 70-180) and questionnaires will be compared from baseline to 6 and 12 months using linear regression procedures as detailed above.

DETAILED DESCRIPTION:
SUMMARY OF STUDY RATIONAL - Our project focuses on two populations; those with type 1 diabetes (T1D) and those with poorly controlled type 2 diabetes (T2D). Telemedicine Monitoring of Adults with Uncontrolled Diabetes Mellitus (Tele-MONITOR DM) is designed to reduce health care disparities in under resourced populations by enhancing existing telehealth visits for individuals with poorly controlled diabetes through continuous glucose monitoring (CGM) with data automatically transmitted to a clinic dashboard to allow for outreach to patients as needed in between routinely scheduled visits and feedback to primary care providers for medication management.

Few people with diabetes reach their treatment targets. This is particularly true for the under resourced who lack access to medical care who often have very high glucose levels, as well as have a risk for hypoglycemia. For our patients, part of the difficulty in accessing care is the disruption it creates in their schedule to take the time to come in for an office visit. The use of telemedicine due to the COVID pandemic has expanded our ability to reach patients in a convenient manner, based on the patient's preferences rather than a fixed clinic schedule. Use of technology has increased along with this, particularly because Medicare rules for covering technology have expanded. This allows for close monitoring and frequent medication dose adjustment to treat both hyper- and hypo-glycemia. These lessons learned during COVID create a new opportunity to expand the use of technology to underserved areas where uptake has been lagging but where the need is greatest.

Our system of monitoring, which the investigators originally called Tele-CGM will send alerts to our clinic that will allow for outreach to patients who need assistance, rather than waiting for them to contact the clinic. By looking both at the daily alerts as well as weekly data updates on each patient, the investigators should help keep patients safer, start and uptitrate guideline-recommended medications more effectively and work to encourage adherence to lifestyle and medications. Originally, the investigators had hoped to develop our Tele-CGM system to include data from all CGM systems. Unfortunately this is not currently possible. Therefore the investigators plan to work the Freestyle Libre 2. The data will be monitored through the existing LibreView system, with enhanced functionality for population management. The CGM system selected for each patient will be individualized based on the patient's preferences, clinical need for the device and insurance coverage (if available). For those without a CGM, they will be provided with a Freestyle Libre device free of charge.

If our findings prove the utility of our system, it will validate the role of treatment intensification for diabetes management in primary care, using asynchronous data collection from CGM devices by diabetes educators supervised by an endocrinologist. It will also assess the utility of a device-dashboard that will provide near real-time alerts to clinic staff so that they can respond to unusually high and low blood glucose values as well as discontinuation of sensor use.

INTERVENTION Baseline Visit-Visit 1 1. Obtain informed consent 2. Obtain clinical data on patient including diabetes and medical history 3. Administer questionnaires 4. Measure point of care HbA1C 5. Start blinded CGM device (even if using their own CGM) Baseline Blinded CGM wear - Visit 2

1. Downloaded from the patient's blinded CGM device.
2. Teach the patient how the remote monitoring systems works.
3. The patient will be signed into the LibreView portal using a research code name and email.
4. Systems will be checked to be sure they are functioning
5. Remote monitoring program will be activated.
6. Telemedicine procedure will be discussed with patient; emergency contact numbers will be obtained in case patient cannot be reached.
7. Telemonitoring will commence (see below)
8. Recommendations will be given to the patient and his/her provider for medication adjustment/intensification following the Los Angeles County Department of Health Services Protocols for Diabetes Management.
9. Patient will be given basic education information and a link to Los Angeles County + University of Southern California patient educational videos. They will be able to watch these videos at home or in clinic.

Month 6 - Blinded CGM Visit 3

1. Provided blinded CGM device (in-person or by mail) three weeks prior to Visit 2
2. Instruct subjects to monitor their glucose levels with the their usual method (CGM or BGM) during the blinded CGM period.

6 Month Visit - Visit 4

1. Administer questionnaires
2. Measure point of care HbA1C
3. Collect blinded CGM data
4. Review and document medication use, hospitalizations/emergency department/outpatient (in-person or telemedicine) visits Month 12 - Blinded CGM

1. Provided blinded CGM device (in-person or by mail) three weeks prior to Visit 2 2. Instruct subjects to monitor their glucose levels with the their usual method (CGM or BGM) during the blinded CGM period.

12 Month Visit - Visit 6

1. Administer questionnaires
2. Measure point of care HbA1C
3. Collect blinded CGM data
4. Review and document medication use, hospitalizations/emergency department/outpatient (in-person or telemedicine) visits DATA COLLECTION AND TESTING PROCEDURES (Baseline, 6 months and 12 months) HbA1c - HbA1c will be obtained using the point of care Siemens DCA Vantage Analyzer.

Continuous Glucose Monitoring (CGM) Blinded Mode - A commercially available Libre Pro (for blinded mode) CGM device will be provided and a sensor will be inserted.

Data from TeleMonitor Program (using FDA approved LibreView), including frequency and types of alerts, action taken. A commercially available Libre 2 CGM device will be provided and a sensor will be inserted. The participant will receive instructions on calibration, insertions, maintenance, use, and removal of the sensor. The Libre 2 CGM is linked to the LibreView program which captures CGM data and initiates alerts based on the following parameters:

1. ≥4 hours without CGM signal
2. ≥2 hours 54 - 70 mg/dl
3. 15 minutes <54 mg/dl Brief Patient Health Questionnaire (PHQ-8) - The PHQ-8 is an eight-item scale developed specifically to screen for depression. Each question has a choice format of the number of days in the past two weeks the question apply to them (Not at all 0-1day, Several days 2-6 days, More than half the days 7- 11 days, and Nearly every day 12-14 days). Administration time is approximately 10 minutes.

Diabetes Treatment Satisfaction Questionnaire (DTSQ) - The DTSQ assess patient satisfaction with diabetes treatment each. It is composed of eight questions, each of which is scored by patients on a scale ranging from zero (e.g., "very dissatisfied", "very inconvenient") to six (e.g., "very satisfied", "very convenient"). The questionnaire is composed of two different factors. The first factor assesses treatment satisfaction and consists of six questions (Q 1, 4, 5, 6, 7 and 8). These six questions ask about "satisfaction with current treatment", "flexibility", "convenience", "understanding of diabetes", "recommend treatment to others" and "willingness to continue", respectively. The second factor consists of two questions (Q 2 and 3), which assess the burden from hyper- and hypoglycemia, respectively (zero being "none of the time" to six being "most of the time"). Treatment satisfaction is assessed as the sum of the scores of the six questions on the first factor (total score 36), with a higher score indicating higher treatment satisfaction. Administration time is approximately 10 minutes.

Glucose Monitoring Satisfaction Survey (GMSS) - The GMSS assess treatment satisfaction with glucose monitoring devices and its impact on quality of life and other patient-reported outcomes for patients with type 1 and type 2 diabetes. It is a 15 item scale asking subjects how much they agree or disagree (Likert scale 1-5) with each statement as it pertains to their current glucose monitor. There are 4 sub-scales Openness, Emotional burden, Behavioral burden, and Trust (for type 1) Worthwhileness (for type 2). Higher scores indicate higher satisfaction. Administration time is approximately 10 minutes.

Diabetes Distress Scale for T1D (DDS T1D) - The DDS T1D is a 28-item self-report scale that highlights seven critical dimensions of distress: powerlessness, management distress, hypoglycemia distress, negative social perceptions, eating distress, physician distress, and friends/family distress. The seven sub-scales include:

Powerlessness: A broad sense of feeling discouraged about diabetes; e.g., "feeling that no matter how hard I try with my diabetes, it will never be |good enough." Management Distress: Disappointment with the patient's self-care efforts; e.g., "feeling that I don't give my diabetes as much attention as I probably should." Hypoglycemia Distress: Concerns about hypoglycemic events; e.g., "feeling that I can't ever be safe from the possibility of a serious hypoglycemic event." Negative Social Perception Distress: Concerns about the possible negative judgments of others; e.g., "feeling like I have to hide my diabetes from other people.

Eating Distress: Concerns that the patient's eating is out of control; e.g., "feeling that thoughts about food and eating control my life." Physician Distress: Disappointment with the patient's current health care professionals; e.g., "feeling that I don't get help I really need from my diabetes doctor about managing diabetes." Friend/Family Distress: A perception that there is too much focus on diabetes amongst the patient's loved ones; e.g., "feeling that my family and friends make a bigger deal out of diabetes than they should." Higher scores indicate higher stress. Administration time is approximately 15 minutes.

Diabetes Distress Scale for T2D (DDS T2D) - The DDS T2D is a 17 item self-report scale that reflects overall diabetes distress from all sources with four sub-scales:

Emotional Burden (5 items): feeling overwhelmed, frightened or fearful about managing the demands of diabetes over time.

Regimen Distress (5 items): feeling that they are failing by not managing their diabetes well, e.g., meal plan, exercise, etc.

Interpersonal Distress (3 items): feeling that they are not receiving sufficient support for their diabetes among family and friends.

Physician Distress (4 items): worries about health care and obtaining sufficient expertise, support and direction from health care providers.

Each question is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem." Higher scores indicate higher stress. Administration time is approximately 10 minutes.

Assessment of Sever Hypoglycemia and Diabetic Ketoacidosis -The Assessment of Severe Hypoglycemia and Diabetic Ketoacidosis is an interviewer administered survey assessing if the subject had any episodes of severe hypoglycemia and/or diabetic ketoacidosis since their last study visit. Events are recorded to assess frequency, as is type of assistance required to treat the event. Administration time is approximately 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 or type 2 diabetes for at least 6 months
2. HbA1C >8% or any episode of level three hypoglycemia or diabetic ketoacidosis (DKA) in the past 6 months or at least once weekly episodes of level 1 or 2 hypoglycemia
3. Age >18 years old
4. On medication for treatment of diabetes-any oral or injectable agents on a stable dose of medication for at least 3 months.
5. If on insulin performing blood glucose monitoring (BGM) at least 3 times per week
6. Patients may be current continuous glucose monitor (CGM) users, prior CGM users or naïve to CGM.
7. No serious illnesses where life expectancy is <1 year
8. Understand the study requirements and agree to comply with all study visits and procedures, including the use of the study CGM.
9. Fluent in English or Spanish
10. Must have a smart phone or access to a computer that can connect to LibreView.
11. Under the care of a Los Angeles County + University of Southern California provider who can prescribe diabetes medications and make dose adjustments/medication intensification as needed.

Exclusion Criteria:

1. Severe tape allergy
2. Visual impairment such that CGM data cannot be viewed.
3. On dialysis
4. History of an adverse reaction to wearing CGM in the past (e.g., increased anxiety and/or an increase in acute diabetes complications such as DKA/severe hypoglycemia).
5. Subject is currently pregnant or lactating or plan on becoming pregnant during the course of the study.
6. Subject cannot follow instructions due to a medical condition or mental illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 English or Spanish speaking subjects (125 adults with type 2 and 75 with type 1 diabetes)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
CGM - Tele-monitoring effects on HbA1c | 12-months
  Number of patients with decreased HbA1c as measured by point of care HbA1c level from baseline to 12 months.

SECONDARY OUTCOMES:
CGM-Tele-monitoring effects on CGM adherence | 12-months
  Number of patients with increased CGM use as assessed by number of days CGM data is available for download from baseline to 12 months
CGM-Tele-monitoring effects on glucose time in range (TIR) | 12-months
  Number of patients with weekly increased percent of time their glucose is in range (TIR; CGM glucose levels between 70-180) as assessed by CGM data download from baseline to 12 months
CGM-Tele-monitoring effects on depression | 12 months
  Number of patients with decreased depression as measured by PHQ 8 from baseline to 12 months.
CGM-Tele-monitoring effects on glucose monitoring satisfaction | 12 months
  Number of patients with increased glucose monitoring satisfaction as measured by GMSS from baseline to 12 months.
CGM-Tele-monitoring effects on diabetes treatment satisfaction | 12 months
  Number of patients with decreased depression as measured by DTSQ from baseline to 12 months.
CGM-Tele-monitoring effects on diabetes treatment satisfaction | 12 months
  Number of patients with increased diabetes treatment satisfaction as measured by DTSQ from baseline to 12 months.
CGM-Tele-monitoring effects on protocol driven enhancement of therapy with Glucagon-Like Peptide-1 Receptor Agonist (GLP-1RA) and sodium-glucose cotransporter -2 (SGLT-2) inhibitors | 12 months
  Number of patients with new prescriptions for GLP-1 RA and SGLT-2 inhibitors from baseline to 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California Eastside Center for Diabetes, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No